CLINICAL TRIAL: NCT02693886
Title: Clinical Study That Effect of Individualized Intervention of Single Colonoscopy on Colorectal Adenomas Detection
Brief Title: Effect of Single Colonoscopy on Colorectal Adenomas Detection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WX0302-B010507-150031-PB
Record Dates: First submitted 2016-01-27; First posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- A group: Experience of endoscopist: >2000 cases
  Interventions: Other: doctor experience
- B group: Experience of endoscopist:between 1000 and 2000 cases
  Interventions: Other: doctor experience
- C group: Experience of endoscopist:between 500 and 1000 cases
  Interventions: Other: doctor experience
- D group: Experience of endoscopist:<500 cases
  Interventions: Other: doctor experience

INTERVENTIONS:
Other: doctor experience

SUMMARY:
Individualized colonoscopy withdrawal time is determined based on the different grade of physician experience and quality of bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than the age of 40;
2. Pathology and endoscopic data recorded available and detailed;
3. Whole bowel staining endoscopy is not done.

Exclusion Criteria:

1. Not reach the ileocecal junction;
2. Colorectal cancer;
3. Familial adenomatous polyposis;
4. Inflammatory bowel disease;
5. Part of the bowel resection.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. greater than the age of 40;
  2. Pathology and endoscopic data recorded available and detailed;
  3. Whole bowel staining endoscopy is not done.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of polyps in different withdraw time | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Detection rate of polyps in different experiment levels of examiners | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Yes